CLINICAL TRIAL: NCT01275729
Title: The Effect of Loop Diuretics on Severity and Outcome of Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-503-B
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Acute Kidney Failure
Keywords: Renal Replacement Therapy; Diuretics; Biomarkers; Renal Insufficiency; Furosemide; Therapeutic Uses; Physiological Effects of Drugs; Biological Markers
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lasix (Experimental): Pt to get dose of furosemide after meeting entry criteria - dose dependent on previous exposure to diuretics
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — dose: 1 mg / kg (iv) if the patient is furosemide naive or 1.5 mg/kg (iv) if the patient is not furosemide naive
  Other Names: Laisx

SUMMARY:
The primary objective is to safely determine if the investigators can identify the severity of Acute Kidney Injury (AKI) early in the course of the disease. Once enrolled the investigators will draw blood and urine for novel and standard biomarkers. The investigators are attempting to determine if these biomarkers can forecast the course of AKI (need for dialysis, death and renal recovery). The investigators seek to determine how well physicians caring for those with AKI can predict the clinical course compared to these novel biomarkers of AKI and if there is an association between clinical course and 3 year patient outcomes.

DETAILED DESCRIPTION:
AKI is a very common disease in the setting of critical illness and carries an extremely high morbidity and mortality rate (over 50%). Currently there are no FDA approved therapeutic agents for the treatment of AKI. There is limited prospective evidence to guide nephrologists in terms of which patients will progress to more severe AKI in the setting of early AKI. Similarly, there is no evidence to guide nephrologists in terms of which patients will completely recover their renal function after AKI. Thus we need to know very early in the course of AKI which patients will progress and go on to require renal replacement therapy (RRT). Additionally we will investigating the long term patient outcomes, 2-3 years after the index AKI admission.

ELIGIBILITY:
Inclusion Criteria:

1. 18 yrs or older
2. increase in serum creatinine of 0.3 mg/dl within 48 hours or an increase of greater than or equal to 150% from baseline or sustained oliguria (UOP < 0.5 cc/kg/hr for 6 hours with the last 48hours)
3. written informed consent
4. patients with an indwelling bladder catheter

Exclusion Criteria:

1. Voluntary refusal
2. Patients with advanced chronic kidney disease - as defined by a baseline glomerular filtration rate (GFR) < 30 ml/min (MDRD)
3. history of renal transplant
4. Pregnant patients
5. Allergy / Sensitivity to Loop diuretics (furosemide)
6. Pre-renal AKI

   * defined by a Fractional Excretion of Sodium (FENa) of < 1% and no urinary casts
   * under-resuscitated as per the treating clinical team
   * active bleed
7. Post renal AKI

   * evidence of hydro-ureter
   * clinical scenario wherein obstruction is considered a likely possibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay L Koyner, MD, Principal Investigator — University of Chicago
Locations (4):
- United States (4):
  - University of California-San Francisco, San Francisco, California
  - George Washington University, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Medicine, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lasix
Started | 96
Completed | 92
Not Completed | 4
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lasix
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (14.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 59
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 42
  Caucasian | 41
  Native | 1
  Other | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression to Stage 3 AKI
Description: The number of patients who progressed to Stage 3 during the time of observation
Time Frame: within 7 days of furosemide administration
Measure: Count of Participants; unit: Participants
Arm/Group | Lasix
Number analyzed (Participants) | 92
Participants | 23

2. Primary Outcome: Receipt of Renal Replacement Therapy (RRT)
Description: The number of patients who received renal replacement therapy (Dialysis)
Time Frame: within 7 days of furosemide administration
Measure: Count of Participants; unit: Participants
Arm/Group | Lasix
Number analyzed (Participants) | 92
Participants | 10

3. Primary Outcome: Death
Description: Inpatient mortality
Time Frame: During the index hospital stay, an average of 17 days, until hospital discharge, or until death, whatever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Lasix
Number analyzed (Participants) | 92
Participants | 16

4. Secondary Outcome: Length of Intensive Care Unit (ICU) Stay
Description: duration if ICU stay for all patients
Time Frame: During the index hospital stay, an average of 9 days, until ICU discharge, or until death, whatever occurs first
Measure: Mean (Standard Error); unit: days
Arm/Group | Lasix
Number analyzed (Participants) | 92
days | 9.15 (1.45)

5. Secondary Outcome: Length of Hospital Stay
Description: duration of the total hospital Stay for all patients
Time Frame: During the index hospital stay, an average of 17 days, until hospital discharge, or until death, whatever occurs first
Measure: Mean (Standard Error); unit: days
Arm/Group | Lasix
Number analyzed (Participants) | 92
days | 17.29 (2.4)

ADVERSE EVENTS:
Time Frame: During the index hospital stay, an average of 17 days, until hospital discharge, or until death, whatever occurs first
Arm/Group | Lasix
All-Cause Mortality (participants affected / at risk) | 16/92
Serious Adverse Events (participants affected / at risk) | 0/92
Other Adverse Events (participants affected / at risk) | 19/92
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lasix (N=92)
Hypotension- defined requiring intervention by means of fluid administration or vasopressor support (Cardiac disorders) | 9
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT01275729/Prot_SAP_000.pdf